CLINICAL TRIAL: NCT03426267
Title: A Randomized, Double-Masked, Parallel Group, Multicenter, Study To Evaluate Efficacy And Safety of SDN -037 Twice Daily Compared With Vehicle For The Treatment Of Inflammation And Pain Associated With Ocular Surgery.
Brief Title: Evaluation of Efficacy and Safety of SDN-037
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLR_16_31
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Results first posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Inflammation and Pain Associated With Ocular Surgery
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SDN-037 (Experimental)
  Interventions: Drug: SDN-037
- vehicle (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SDN-037 — twice daily
  Arms: SDN-037
Drug: Placebo — twice daily
  Arms: vehicle

SUMMARY:
The efficacy and safety of SDN-037 twice daily will be evaluated and compared with vehicle for the treatment of inflammation and pain associated with ocular surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 2 years of age on the date of assent or 18 years of age at the date of consent
2. Be able and willing to follow study instructions and complete all required visits
3. Females of childbearing potential must not be pregnant (as confirmed by a negative urine pregnancy test
4. Able to self-instill the IP or have a caregiver available to instil all doses of the IP

Exclusion Criteria:

1. Any known allergy or hypersensitivity to difluprednate therapy
2. An acute ocular infection (bacterial, viral or fungal) or active ocular inflammation in the study eye
3. Any active corneal pathology noted in the study eye
4. Currently suffering from alcohol and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - SPARC Site 13, Chandler, Arizona
  - SPARC Site 14, Mesa, Arizona
  - SPARC Site 11, Prescott, Arizona
  - SPARC Site 12, Sun City, Arizona
  - SPARC site 01, Fayetteville, Arkansas
  - SPARC Site 10, Santa Barbara, California
  - SPARC Site 08, Colorado Springs, Colorado
  - SPARC Site 06, Coral Springs, Florida
  - SPARC Site 18, Fort Myers, Florida
  - SPARC Site 16, Jacksonville, Florida
  - SPARC Site 07, Miami, Florida
  - SPARC Site 15, Paducah, Kentucky
  - SPARC Site 05, Saint Joseph, Michigan
  - SPARC Site 09, Henderson, Nevada
  - SPARC Site 03, Poughkeepsie, New York
  - SPARC Site 04, Winston-Salem, North Carolina
  - SPARC Site 17, Fargo, North Dakota
  - SPARC Site 19, Austin, Texas
  - SPARC Site 2, Mission, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SDN-037: dosage: SDN-037
  dosage form: solution
  frequency of administration: twice daily
- Vehicle: dosage: Placebo
  dosage form: solution
  frequency of administration: twice daily
Period: Overall Study
Arm/Group | SDN-037 | Vehicle
Started | 163 | 162
Modified Intent-to-Treat Population | 154 | 144
Completed | 142 | 90
Not Completed | 21 | 72
Not completed — Physician Decision | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Protocol Violation | 1 | 3
Not completed — Adverse Event | 9 | 27
Not completed — Prohibited Treatment Intake | 2 | 3
Not completed — Lack of Efficacy | 0 | 25
Not completed — other | 3 | 0

BASELINE CHARACTERISTICS:
Population: modified intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | SDN-037 | Vehicle | Total
Number analyzed (Participants) | 154 | 144 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (8.61) | 68.3 (8.94) | 68.3 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 84 | 178
  Male | 60 | 60 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 42 | 81
  Not Hispanic or Latino | 114 | 102 | 216
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 31 | 65
  White | 115 | 109 | 224
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Subjects With an Anterior Chamber Cell Grade of 0 at Day 15
Description: Grade Cell Count 0 0
  1. 1-10
  2. 11-20
  3. 21-50
  4. > 50
  ACC grade of 0 at the Day 15 visit was considered a responder to therapy ACC score of >0 at Day 15 visit was considered a failure (or non-responder)
Time Frame: Day 15
Population: Modified Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | SDN-037 | Vehicle
Number analyzed (Participants) | 154 | 144
Participants | 96 | 30
Statistical Analysis 1: Comparison: SDN-037 vs Vehicle; Test type: Other; p < .0001, Chi-squared

2. Secondary Outcome: Subjects Who Achieve a Pain Score of 0 at Day 15
Description: Pain was assessed using a visual analog scale (VAS). The Visual Analog Scale (VAS) uses a 100 mm (10 cm) line (0 = absent >100 = maximum). A 0 indicates an absence of pain A higher score indicates greater pain intensity.
Time Frame: Day 15
Population: Modified Intent-To-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | SDN-037 | Vehicle
Number analyzed (Participants) | 154 | 144
Participants | 151 | 106
Statistical Analysis 1: Comparison: SDN-037 vs Vehicle; Test type: Other; p < .0001, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 6 visits over a period of 22 to 36 days
Arm/Group | SDN-037 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/144
Serious Adverse Events (participants affected / at risk) | 2/154 | 2/144
Other Adverse Events (participants affected / at risk) | 87/154 | 96/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SDN-037 (N=154) | Vehicle (N=144)
Rhegmatogenous Retinal Detachment In Study Eye (Eye disorders) | 0 (0) | 1 (1)
Left Foot Infection Secondary To Trauma (Infections and infestations) | 1 (1) | 0 (0)
Cystoid Macula Edema (Eye disorders) | 1 (2) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SDN-037 (N=154) | Vehicle (N=144)
Anterior chamber cell (Eye disorders) | 26 (87) | 35 (96)
Anterior chamber flare (Eye disorders) | 15 (87) | 31 (96)
Visual acuity reduced (Eye disorders) | 14 (87) | 30 (96)
Conjunctival hyperaemia (Eye disorders) | 5 (87) | 22 (96)
Corneal oedema (Eye disorders) | 6 (87) | 20 (96)
Eye pain (Eye disorders) | 10 (87) | 14 (96)
Photophobia (Eye disorders) | 6 (87) | 10 (96)
Intraocular pressure increased (Investigations) | 17 (87) | 7 (96)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT03426267/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT03426267/SAP_001.pdf